CLINICAL TRIAL: NCT00921869
Title: A Phase I Dose-finding Study of E7050 Administered Orally to Patients With Advanced Solid Tumors.
Brief Title: A Study of E7050 Administered Orally to Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7050-J081-102
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Solid Tumors
Keywords: Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms | interventions — N-(2-fluoro-4-((2-(4-(4-methylpiperazin-1-yl)piperidin-1-yl)carbonylaminopyridin-4-yl)oxy)phenyl)-N'-(4-fluorophenyl)cyclopropane-1,1-dicarboxamide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7050

INTERVENTIONS:
Drug: E7050 — The starting dose of E7050 will be 50 mg given orally, twice-daily, in patients with advanced tumors that have progressed following effective therapy.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD), safety, pharmacokinetics (PK), pharmacodynamics (PD) and anti-tumor activity of E7050 when administered orally twice daily to patients with advanced solid tumors.

DETAILED DESCRIPTION:
Phase I, open-label, dose-escalation study to determine the maximum tolerated dose (MTD) of E7050 given orally, twice-daily, in patients with advanced tumors that have progressed following effective therapy.

ELIGIBILITY:
Inclusion criteria:

1. Subjects with a histological or cytological diagnosis of solid tumors or gastric cancer.
2. Subjects who have progressed after treatment with approved therapies or for whom there are no standard effective therapies available.
3. Subjects with adequate organ function.
4. Patients who have no carryover of effect from prior therapy or no adverse drug reactions (excluding alopecia) that may affect the safety evaluation of the investigational drug.
5. Subjects with Performance Status (PS) 0-1 established by Eastern Cooperative Oncology Group (ECOG).

Exclusion criteria:

1. Subjects who have brain metastases with clinical symptoms or which requires treatment.
2. Subjects with the serious complications or disease history.
3. Subjects who cannot take oral medication.
4. Subjects who need continuous use of drugs or foods that strongly inhibit or induce CYP3A4/5 or CYP2D6 during the study period.
5. Female subjects who are pregnant or breast-feeding.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determination of the MTD of E7050 given orally twice daily. MTD is the highest dose at which no more than 1 out of 6 patients experiences dose-limiting toxicity (DLT) | During the Run-in Phase and the first 5 weeks of treatment

SECONDARY OUTCOMES:
Dose-limiting toxicities. | During the Run-in Phase and the first 5 weeks of treatment
Incidence and severity of adverse events and their drug relationship. | Throughout the entire study
PK of blood and urine | During the Run-in Phase, Cycle 1 (28 days) and Day 15 of Cycle 2 for blood; Day 28 of Cycle 1 for urine
Pharmacodynamic (PD) biomarker analysis of blood and tumor tissue samples. | During Cycle 1 (28 days) and Day 15 of Cycle 2 for blood; on Day 22 of Cycle 1 for optional tumor biopsies
Best overall tumor response, duration of response and stable disease, assessed by Response Evaluation Criteria in Solid Tumors. | Every 4 weeks for complete and partial response; by 7th week for stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Sawada, Study Director — Oncology Clinical Development Section. JAC PCU. Eisai Co., Ltd.
Locations (1):
- Kashiwa-shi, Chiba, Japan